CLINICAL TRIAL: NCT00804492
Title: Bureau of Health Promotion,Department of Health, R.O.C. (Taiwan)
Brief Title: Establishment of an Integrated Model for Prevention of Elderly Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jau-Yih Tsauo, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200710010R
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Falls
Keywords: To organize a multidisciplinary team for integrated falls prevention; To draft a guideline for falls prevention in the elderly; To set up a multidisciplinary fall clinic; To set up a falls prevention classroom; To enhance cooperate between hospitals and primary care units for falls prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): To establish an integrated intervention model for prevention of elderly fall
  Interventions: Behavioral: Multifaceted intervention
- 2 (Experimental): To perform a RCT to investigate the effectiveness of the multicenter, multifaceted intervention program
  Interventions: Behavioral: Multifaceted intervention

INTERVENTIONS:
Behavioral: Multifaceted intervention — consulted, educated, referred or receive an exercise training for their fitness, strength and balance

SUMMARY:
Falls, with a high prevalence, high risk and consequent medical and social costs, are an important issue for medical care and health promotion in the elderly. The prevalence of falls in the elderly lies in between 10-20%. Falls have become the second leading cause of death from injury for the elderly in Taiwan. A community-based study showed that, among those old adults after a fall, 27.3% were severely injured, 53.9% got a minor injury, and only 18.9% remained intact. Another study revealed that among fall injury events reported, 42% were hospitalized, of whom 2.2% died in hospital, and 37% entered nursing homes after discharge from hospital. In addition to physical discomfort, half of the elderly fallers would become disabled, and bring a heavy burden of social economy and family care. It was estimated that there were 460 thousand of old people who had a fall, and 125 thousand of them were injured in Taiwan, 2007. Research evidence shows that falls prevention is effective and feasible. Although primary falls prevention programs have been conducted at the community level and extended to 25 counties and cities for many years, they were not integrated with secondary and tertiary prevention. The study aims to establish an integrated fall prevention model, combined with primary, secondary and tertiary prevention. The model will be practiced in participating hospitals and communities, with a randomized control trial (RCT) design to examine its feasibility and effectiveness. Our study subjects are persons aged 65 and over who live in communities, go to out-patient departments (OPD) or emergency room (ER) care.

Tasks for implementation

1. To organize a multidisciplinary team for integrated falls prevention.
2. To draft a guideline for falls prevention in the elderly.
3. To set up a multidisciplinary fall clinic.
4. To set up a falls prevention classroom.
5. To enhance cooperate between hospitals and primary care units to fulfill the guideline for falls prevention in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Old people (65 years old or more)
* With at least one fall in the past one year, or with disease related to fall, such as central nerve system disease or lower extrimity fracture

Exclusion Criteria:

* The result of screening test is "no fall risk"
* Cannot be followed for 6 months
* Cannot be evaluated because of the mental status
* Cannot have the exercise intervention
* Falling due to expected reason, such as suffering heart atteck

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The number and severity of fall | once per month for 6 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Jau-Yih Tsauo, Taipei, Taiwan, Taiwan